CLINICAL TRIAL: NCT00910104
Title: Cholestasis Reversal: Efficacy of IV Fish Oil
Acronym: Reversal
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mark Puder (Other)
Responsible Party: Sponsor-Investigator, Mark Puder, M.D., Ph.D, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-04-048; 1R01FD003460-02 (FDA)
Record Dates: First submitted 2009-05-20; First posted 2009-05-29 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Parenteral Nutrition Associated Liver Disease; Short Bowel Syndrome; Gastrointestinal Disease
Keywords: PNALD; Omegaven; Parenteral Nutrition Associated Liver Disease; Cholestasis; Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome; Gastrointestinal Diseases; Cholestasis | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omegaven (Experimental): 1g/kg/day for duration of study participation for all participants
  Interventions: Drug: Omegaven®

INTERVENTIONS:
Drug: Omegaven® — 10% Omegaven® 1g/kg/day, IV (in the vein) until the patient no longer requires parenteral nutrition or until participation in the study is terminated
  Other Names: Fish Oil Lipid Emulsion (FOLE)

SUMMARY:
The purpose of this study is to determine whether Omegaven is effective in the treatment of parenteral nutrition associated liver disease (PNALD).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the omega-3 fatty acid emulsion (Omegaven), when used in lieu of the conventional soy-based fat emulsion (Intralipid), is effective in the treatment of parenteral nutrition associated liver disease (PNALD).

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be PN dependent (unable to meet nutritional needs solely by enteral nutrition) and are expected to require PN for at least another 30 days
2. Patients considered eligible for study participation must have parenteral nutrition associated liver disease (PNALD) as defined as a direct bilirubin of > 2 mg/dl or currently on Omegaven through another protocol. Other causes of liver disease should be excluded. A liver biopsy is not necessary for treatment.
3. Direct bilirubin > 2.0 mg/dl or already on Omegaven through another protocol
4. Signed patient informed consent.
5. The patient must have utilized standard therapies to prevent the progression of his/her liver disease including surgical treatment, cyclic PN, avoiding overfeeding, reduction/removal of copper and manganese from PN, advancement of enteral feeding, and the use of ursodiol (i..e., Actigall®).

Exclusion Criteria:

1. Pregnancy
2. Other causes of chronic liver disease (Hepatitis C, biliary atresia, and alpha 1 anti-trypsin deficiency).
3. Enrollment in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team)
4. The parent or guardian or child unwilling to provide consent or assent

In rare instances, patients diagnosed with PNALD may later be found to have liver disease due to other causes in addition to the use of PN (i.e., inborn errors of metabolism, viral infections ). Such causes may not be known at the time of enrollment and will not preclude them from continuing in the study. For the sake of statistical analysis, however, these patients will be excluded although all data will be collected and reviewed.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gura KM, Lee S, Valim C, Zhou J, Kim S, Modi BP, Arsenault DA, Strijbosch RA, Lopes S, Duggan C, Puder M. Safety and efficacy of a fish-oil-based fat emulsion in the treatment of parenteral nutrition-associated liver disease. Pediatrics. 2008 Mar;121(3):e678-86. doi: 10.1542/peds.2007-2248. PMID 18310188
- [Background] Gura KM, Duggan CP, Collier SB, Jennings RW, Folkman J, Bistrian BR, Puder M. Reversal of parenteral nutrition-associated liver disease in two infants with short bowel syndrome using parenteral fish oil: implications for future management. Pediatrics. 2006 Jul;118(1):e197-201. doi: 10.1542/peds.2005-2662. PMID 16818533
- [Background] Nandivada P, Anez-Bustillos L, O'Loughlin AA, Mitchell PD, Baker MA, Dao DT, Fell GL, Potemkin AK, Gura KM, Neufeld EJ, Puder M. Risk of post-procedural bleeding in children on intravenous fish oil. Am J Surg. 2017 Oct;214(4):733-737. doi: 10.1016/j.amjsurg.2016.10.026. Epub 2016 Dec 1. PMID 27979360
- [Background] Nandivada P, Baker MA, Mitchell PD, O'Loughlin AA, Potemkin AK, Anez-Bustillos L, Carlson SJ, Dao DT, Fell GL, Gura KM, Puder M. Predictors of failure of fish-oil therapy for intestinal failure-associated liver disease in children. Am J Clin Nutr. 2016 Sep;104(3):663-70. doi: 10.3945/ajcn.116.137083. Epub 2016 Aug 10. PMID 27510535
- [Background] Nandivada P, Fell GL, Mitchell PD, Potemkin AK, O'Loughlin AA, Gura KM, Puder M. Long-Term Fish Oil Lipid Emulsion Use in Children With Intestinal Failure-Associated Liver Disease [Formula: see text]. JPEN J Parenter Enteral Nutr. 2017 Aug;41(6):930-937. doi: 10.1177/0148607116633796. Epub 2016 Mar 9. PMID 26962059
- [Background] Nandivada P, Chang MI, Potemkin AK, Carlson SJ, Cowan E, O'loughlin AA, Mitchell PD, Gura KM, Puder M. The natural history of cirrhosis from parenteral nutrition-associated liver disease after resolution of cholestasis with parenteral fish oil therapy. Ann Surg. 2015 Jan;261(1):172-9. doi: 10.1097/SLA.0000000000000445. PMID 24374535
- [Background] Le HD, de Meijer VE, Robinson EM, Zurakowski D, Potemkin AK, Arsenault DA, Fallon EM, Malkan A, Bistrian BR, Gura KM, Puder M. Parenteral fish-oil-based lipid emulsion improves fatty acid profiles and lipids in parenteral nutrition-dependent children. Am J Clin Nutr. 2011 Sep;94(3):749-58. doi: 10.3945/ajcn.110.008557. Epub 2011 Jul 20. PMID 21775562
- [Result] Puder M, Valim C, Meisel JA, Le HD, de Meijer VE, Robinson EM, Zhou J, Duggan C, Gura KM. Parenteral fish oil improves outcomes in patients with parenteral nutrition-associated liver injury. Ann Surg. 2009 Sep;250(3):395-402. doi: 10.1097/SLA.0b013e3181b36657. PMID 19661785
- [Derived] Gura KM, Calkins KL, Premkumar MH, Puder M. Use of Intravenous Soybean and Fish Oil Emulsions in Pediatric Intestinal Failure-Associated Liver Disease: A Multicenter Integrated Analysis Report on Extrahepatic Adverse Events. J Pediatr. 2022 Feb;241:173-180.e1. doi: 10.1016/j.jpeds.2021.10.030. Epub 2021 Oct 23. PMID 34695449
- [Derived] Gura KM, Premkumar MH, Calkins KL, Puder M. Fish Oil Emulsion Reduces Liver Injury and Liver Transplantation in Children with Intestinal Failure-Associated Liver Disease: A Multicenter Integrated Study. J Pediatr. 2021 Mar;230:46-54.e2. doi: 10.1016/j.jpeds.2020.09.068. Epub 2020 Oct 8. PMID 33038344
- [Derived] Gura K, Premkumar MH, Calkins KL, Puder M. Intravenous Fish Oil Monotherapy as a Source of Calories and Fatty Acids Promotes Age-Appropriate Growth in Pediatric Patients with Intestinal Failure-Associated Liver Disease. J Pediatr. 2020 Apr;219:98-105.e4. doi: 10.1016/j.jpeds.2019.12.065. Epub 2020 Feb 12. PMID 32059815

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2006 and November 2007, 42 patients with IFALD were prospectively enrolled to receive compassionate use open label treatment with 10% FOLE (Omegaven®) as part of their PN. For comparison, retrospective data were retrieved for 49 historical control patients who had received 20% SOLE (Intralipid® 20%) as part of their PN between 1999 and 2006. Patients in both treatment arms were required to have a direct bilirubin level >=2mg/dL upon initiation of their respective lipid emulsion.
Groups:
- Intralipid: Intralipid®: 20% Intralipid® up to 3g/kg/day, IV (in the vein).
Period: Overall Study
Arm/Group | Omegaven | Intralipid
Started | 42 | 49
Completed | 42 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes subjects treated with Omegaven and subjects who served as historical controls treated with Intralipid. Four participants who were transferred to Boston Children's after starting Omegaven at another institution do not have a baseline direct bilirubin (DB). These same four subjects plus two subjects on Intralipid do not have a PN start date, so duration of PN will be unknown in these cases. Therefore, the sample size for DB will be 38+49=87 and for duration of PN 38+47=85.
Groups:
- Intralipid (Historical Control): Patients who received Intralipid between 1999-2006 and whose direct bilirubin was ever >=2.0 mg/dL.
- Total: Total of all reporting groups
Arm/Group | Omegaven | Intralipid (Historical Control) | Total
Number analyzed (Participants) | 42 | 49 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 49 | 91
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 28 | 31 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race and ethnicity not reliably obtained on all subjects.
  Participants
    Hispanic or Latino | 8 | 1 | 9
    Not Hispanic or Latino | 33 | 34 | 67
    Unknown or Not Reported | 1 | 14 | 15
Direct bilirubin [Median (Inter-Quartile Range); unit: mg/dL] — Population: Patients who were transferred to Boston Children's after starting Omegaven elsewhere do not have a baseline direct bilirubin available.
  mg/dL
    number analyzed (Participants) | 38 | 49 | 87
    (all) | 5.5 [3.7 to 8.5] | 3.3 [2.9 to 4.4] | 3.9 [3.1 to 7.0]
Duration of PN before enrollment (d), median (IQR) [Median (Inter-Quartile Range); unit: Days] — Population: PN start date is unknown for n=4 in the fish oil-emulsion arm and n=2 in the soybean oil-emulsion arm.
  Days
    number analyzed (Participants) | 38 | 47 | 85
    (all) | 63 [48 to 118] | 40 [21 to 74] | 54 [33 to 90]

OUTCOME MEASURES:

1. Primary Outcome: Reversal of Cholestasis, Defined as a Direct Bilirubin to <= 2.0 mg/dL.
Description: Time to reversal of established parenteral nutrition associated liver disease, defined as a decrease in direct bilirubin to <= 2.0 mg/dL.
Time Frame: Duration of treatment
Population: The primary efficacy end-point was time to reversal of cholestasis (direct bilirubin <= 2.0 mg/dL).
Measure: Median (Inter-Quartile Range); unit: Weeks
Groups:
- Intralipid (Historical Control): Patients who received Intralipid between 1999 and 2006 and whose direct bilirubin was ever >=2.0 mg/dL.
Arm/Group | Omegaven | Intralipid (Historical Control)
Number analyzed (Participants) | 42 | 49
Weeks | 11.7 [7.7 to 13.9] | 6.4 [3.1 to 9.7]
Statistical Analysis 1: Comparison: Omegaven vs Intralipid (Historical Control); The primary efficacy end-point was time to reversal of cholestasis (direct bilirubin [DB]<=2 mg/dL). Crude (unadjusted) hazard ratios were estimated using proportional hazard regression. Subjects who died, were transplanted, or still on PN at the end of follow-up were censored (Ref: PMID 19661785); Test type: Superiority; p = 0.001, Regression, Cox — All P-values were 2-sided. Analyses were performed in SAS 9.1 (SAS Institute, USA) and S-plus 8 (Insightful, USA). P<0.05 was established as an a priori threshold for statistical significance; Hazard Ratio (HR) = 8.6, 95% CI 2-sided [2.0 to 37.3]
Statistical Analysis 2: Comparison: Omegaven vs Intralipid (Historical Control); The primary efficacy end-point was time to reversal of cholestasis (direct bilirubin [DB]<=2 mg/dL). Adjusted hazard ratios were estimated using proportional hazard regression adjusted for baseline covariates (including duration of parenteral nutrition (PN) and baseline DB). Subjects who died, were transplanted, or still on PN at the end of follow-up were censored (Ref: PMID 19661785); Test type: Superiority; p = 0.001, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 17.4, 95% CI 2-sided [3.7 to 83]
Statistical Analysis 3: Comparison: Omegaven vs Intralipid (Historical Control); Comparison of proportion with reversal of cholestasis (direct bilirubin <=2.0 mg/dL); Test type: Other; p < 0.0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: Safety assessment was made from baseline (start of oil-lipid emulsion) until week 38, at which point only one fish oil-lipid emulsion subject was being followed.
Description: Safety assessment was based on comparison of triglycerides (TG), international normalization ratio (INR), and triene-to-tetraene (T/T) ratio. Hypertriglyceridemia was defined as TG>400 mg/dL, while INR > 2 and T/T ratio > 0.2 were deemed abnormally high.
Groups:
- Omegaven: 1g/kg/day for duration of study participation for all participants
  Omegaven®: 10% Omegaven® 1g/kg/day, IV (in the vein) until the patient no longer requires parenteral nutrition or until participation in the study is terminated
  Please refer to NDA report that summarizes all adverse events reported to FDA
- Intralipid: Soybean oil-lipid emulsion, the standard of care lipid emulsion, with fat doses ranging from 1 to 4 g/kg/d.
Arm/Group | Omegaven | Intralipid
All-Cause Mortality (participants affected / at risk) | 3/42 | 12/49
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/49
Other Adverse Events (participants affected / at risk) | 7/42 | 17/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omegaven (N=42) | Intralipid (N=49)
Hypertriglyceridemia (Investigations) | 2 (2) | 12 (56) — Triglycerides > 400 mg/dL
INR > 2.0 (Investigations) | 3 (9) | 5 (24) — International normalized ratio > 2.0
Essential fatty acid deficiency (Investigations) | 2 (3) | 0 (0) — Triene:tetraene ratio > 0.2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT00910104/Prot_SAP_000.pdf